CLINICAL TRIAL: NCT07019922
Title: A Randomized, Multi-Center, Double-Blind, Sham-Procedure-Controlled Clinical Trial to Investigate the Efficacy and Safety of Elsunersen in Pediatric Participants With Early Onset SCN2A Developmental and Epileptic Encephalopathy
Brief Title: A Clinical Trial of Elsunersen in Pediatric SCN2A-DEE to Assess Efficacy and Safety
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-222-311
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Epileptic Encephalopathy; SCN2A Encephalopathy
Keywords: epilepsis; early onset scn2a; epileptic encephalopathy; scn2a; gain of function; seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: Specific milestones have to be met in Cohort 1 for enrollment to open in Cohort 2 and the same will apply to open Cohort 3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort 1 is the only masked cohort (40 participants). Cohort 2 and Cohort 3 are both open-label and will have 5 participants each.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Arm 1: Double-Blind Treatment Period (Experimental): Double-blind treatment period elsunersen
  Interventions: Drug: 1mg elsunersen
- Cohort 1 Arm 2: Double-Blind Treatment Period (Sham Comparator): Double-blind sham-procedure
  Interventions: Procedure: sham procedure
- Cohort 2: Open-Label Treatment Period (Experimental): Open-label elsunersen
  Interventions: Drug: 1mg elsunersen
- Cohort 3: Open-Label Treatment Period (Experimental): Open-label elsunersen
  Interventions: Drug: 0.5mg elsunersen

INTERVENTIONS:
Drug: 1mg elsunersen — 24 weeks every 4 weeks intrathecally
  Arms: Cohort 1 Arm 1: Double-Blind Treatment Period; Cohort 2: Open-Label Treatment Period
Procedure: sham procedure — 24 weeks of sham-procedure every 4 weeks
  Arms: Cohort 1 Arm 2: Double-Blind Treatment Period
Drug: 0.5mg elsunersen — 24 weeks every 4 weeks intrathecally
  Arms: Cohort 3: Open-Label Treatment Period

SUMMARY:
A Randomized, Multi-Center, Double-Blind, Sham-Procedure-Controlled Clinical Trial to Investigate the Efficacy and Safety of Elsunersen in Pediatric Participants with Early Onset SCN2A Developmental and Epileptic Encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* Has a documented Gain of Function SCN2A variant confirmed through genetic testing.
* Has onset of seizures prior to 3 months of age.
* Seizure frequency of 4 or more countable motor seizures per 28-day during the Baseline Observation Period.

Exclusion Criteria:

* Has any clinically significant or known pathogenic genetic variant other than in the SCN2A gene, or a genetic variant that may explain or contribute to the participant's epilepsy and/or developmental disorder.
* Has bone, spine (eg, kyphosis, scoliosis), bleeding, or other disorder.
* Has received any experimental or investigational drug, device, or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening, including any prior use of gene therapy.
* Is currently pregnant or breastfeeding or is planning to become pregnant during the clinical trial.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of elsunersen on seizure frequency in participants with early-onset SCN2A DEE | 24 weeks
  Median percent change in monthly (28 days) motor seizure frequency from baseline to treatment after 24 weeks

SECONDARY OUTCOMES:
To assess secondary efficacy outcomes of elsunersen in participants with early-onset SCN2A DEE | 24 weeks
  Responder rate - defined as a ≥50% reduction in monthly seizure frequency from baseline compared to treatment after 24 weeks
To assess secondary efficacy outcomes of elsunersen in participants with early-onset SCN2A DEE | 24 weeks
  Change in motor seizure-free days from baseline
CGI-S change from baseline | 24 weeks
  CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use his/her total clinical experience with this patient population and rate the current severity on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
CGI subdomain scores at each postdose time point | 24 weeks
  Clinical Global Impression-Improvement (CGI-I) subdomains scores at each postdose time point
CgGI-S from baseline | 24 weeks
  Caregiver Global Impression-Severity (CgGI-S) at baseline compared to treatment after 24 weeks
CgGI-I subdomain scores at each postdose time point | 24 weeks
  Caregiver Global Impression-Improvement (CgGI I) subdomains scores at each postdose time point
Sleep assessment scores from baseline | 24 weeks
  Sleep assessment scores at baseline compared to each postdose time point
To evaluate the safety and tolerability of elsunersen in participants with early-onset SCN2A DEE | 24 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (2):
- United States (2):
  - Praxis Research Site, San Diego, California
  - Praxis Research Site, Chicago, Illinois